CLINICAL TRIAL: NCT02756169
Title: Effect of an Immediate-postpartum Support by IBCLC to Women With Obesity, on Breastfeeding Performance: A Randomized Trial.
Brief Title: Maternal Obesity and Breastfeeding Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Iberoamericana A.C., Mexico (Other)
Collaborators: Mexican National Institute of Public Health (Other Government); National Council of Science and Technology, Mexico (Other)
Responsible Party: Principal Investigator, Sonia L. Hernandez Cordero, Professor, Universidad Iberoamericana A.C., Mexico
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: SALUD-2014-01-234065; SSA.SEDESA:101/010/01/16 (Other: Ministry of Health of Mexico)
Record Dates: First submitted 2016-04-08; First posted 2016-04-29 (Estimated); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Breastfeeding
Keywords: Obesity; Breastfeeding; Grow up; Milk composition; Mexico
MeSH Terms: conditions — Breast Feeding; Obesity | interventions — Methods

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): One workshop during pregnancy Support for breastfeeding at immediate postpartum Telephonic support after delivery
  Interventions: Other: Intervention
- Control (No Intervention): Standar procedures of neonatal and pregnancy health care at the clinics or hospitals.

INTERVENTIONS:
Other: Intervention — Three actions since pregnancy until the first year of life of the baby for helping the women with obesity to increase the probability of a successful breastfeeding.
  Arms: Intervention

SUMMARY:
Investigators propose this study in order to answer the following research question: An educational intervention and breastfeeding support at postpartum will increase the frequency and total breastfeeding duration in the intervention group? This is a randomized (with control and intervention groups) study, open and parallel (1: 1 ratio between study groups) with 200 pregnant women in the second or third trimester, according to their body mass index (BMI, kg / m2) with excess weight (BMI> 29 pre-pregnancy weight) and that will address their pregnancy in the public health services and hospitals belonging to the Health Ministry of 5 districts: Coyoacán, Magdalena Contreras, Tlalpan, Xochimilco and Alvaro Obregón in Mexico City.

The intervention group and the control group will have the same characteristics for eligibility.

The main phases to develop the study are PHASE 1. INTERVENTION DESIGN PHASE 2. IMPLEMENTATION OF THE INTERVENTION. PHASE 3. FOLLOW-UP The intervention will be offered at 3 times: 1) Educational intervention (a workshop) to pregnant obese women. The workshop will be held by an International Board Certified Lactation Consultant (IBCLC) to promote exclusive breastfeeding and to encourage a better breastfeeding performance in accordance with the WHO recommendations. The workshop will be held at convenient times and will be conducted for groups of 8 to 10 participants; 2) Immediate breastfeeding support at hospital by an IBCLC and; 3) The women will be exposed to early telephonic follow-up during the first week of their children´s lives and each month until six months of life. Then, if the breastfeeding continues, every two months until the first year of their children´s life.

At the first month postpartum, investigators will visit participants at home, both the control group and the intervention group, for collecting information on breastfeeding practices, for taking a breast milk sample to estimate its fatty acids content, and a blood sample (serum) to obtain the C-Reactive Protein. Also, the investigators will take anthropometric measurements of the children to evaluate their growth (weight, length, and skinfold thickness). Investigators will ask for breastfeeding practices and diet of the participants through a 24 hours recall.

The results of this intervention group will be compared with the control group: pregnant obese women without educational intervention or telephonic follow-up.

DETAILED DESCRIPTION:
BACKGROUND Maternal obesity alters the composition of the breast milk beyond the influence of diet on it. Obesity delays copious production of breast milk (Lactogenesis stage II) and it concurs with the synthesis of prolactin (PRL), in response to the decreased sucking of the child.

Besides that, obese mothers have a higher risk of complications in the delivery; where it is common to experience great physiological stress and having a high probability of cesarean, which metabolically does not interfere with breastfeeding but delays its establishment. The excess of subcutaneous fat in the area of the areola of mothers with obesity cause discomfort and stress in the mother and crying in the infant, hindering the correct latch of the infant to the nipple, weakening the neurological stimulus that triggers Prolactin production.

Also, obese mothers have reported an increased feeling of insufficient milk, compared with non-obese mothers and, women with obesity report lower self-efficacy than their pairs without obesity.

Despite the implementation of educational interventions to promote the establishment of breastfeeding in obese women, the results have not been favorable to increase the prevalence of breastfeeding.

To help to improve this practice in women with obesity, it raises the following research question:

An intervention specifically designed to lessen the problems in establishing breastfeeding in women with obesity, which includes: an educational intervention with support during the pregnancy, the immediate postpartum period and the first year of life; increases the frequency of exclusive and predominant breastfeeding during the first month of life, and the total duration of breastfeeding?

METHODOLOGY PHASE 1 INTERVENTION DESIGN The intervention will be made with information derived from a focus group (FG). The main objective is to identify the barriers of a mother with obesity for breastfeeding and, to explore the ideas to overcome them. Investigators will develop a guide to lead the FG discussion.

The main characteristic of women participating in the FG is pregnant women with obesity, the distinction between primiparous and not primiparous women and those who have breastfed before at least for 6 months.

Workshop Design.

With an expert on learning techniques as a collaborator, investigators will design the workshop with the validated messages derived from the FG and it will be complemented by using the experience of an International Board Certified Lactation Consultant (IBCLC). The workshop will be divided into three stages:

* First stage: Basics of breastfeeding and its significance for the health of the baby and mother.
* Second stage: discussion of the problems that may arise, particularly in mothers with obesity. Recommendations and appropriate techniques to solve these problems will be given trough Games and communication activities will be driven.
* Third stage: Treatment of the most common problems and the counseling for solving them.

PHASE 2. IMPLEMENTATION OF THE INTERVENTION. Step 1. Enrollment. This stage is scheduled to take place within 5 months and it has two strategies: 1) with previous authorization of the Health Ministry of Mexico City, investigators will request information from the censuses of each health jurisdiction where there are all the pregnant women identified, or; 2) investigators will approach to pregnant women at the time they attend to their medical consultation.

Once investigators have identified the pregnant women, they will ask for the pregnant women informed consent (adult) / written assent (adolescent) to obtain information about them since the eligibility criteria will be evaluated.

Sociodemographic data and a self-efficacy on breastfeeding questionnaire will be collected. Then, investigators will assign randomly each one of the women to a study group (intervention group or control group).

Step 2. Basal phase. The assignment to a study group is the beginning of the intervention and it is considered as the baseline of the study.

<Activities for the Intervention group>

The intervention will be set at different times:

1. During pregnancy: The workshop. Also, there will be collected another self-efficacy questionnaire at the end.
2. At immediate postpartum: Investigators will identify the arrival of a woman of the study to any of the five hospitals selected for the study. For the intervention group, in addition to the collection of data of health conditions of the mother and her baby, one of the IBCLC will attend and provide immediate support for the establishment of breastfeeding within the first few hours old of the baby. The IBCLC may solve all doubts of the mothers; give support, supervise and guide the initiation of breastfeeding, explain the proper grip, suggest the ideal positions to breastfeeding for both the mother and the newborn, this support it is supposed to be intensive. All these activities must be coordinated with the physicians and nurses from each of the five hospitals in order to follow the rules and requirements that each hospital has established.
3. After delivery and until the first year of life of the children: the intervention will consist of two steps.

   1. During the first 7 days of the life of the infant. An IBCLC will call the mother daily.
   2. A telephonic follow-up at 2 weeks old of the baby and then, a phone call each month until reaching 6 months; then, every two months until the baby will have one year of life. With the calls, investigators pretend to collect information about the duration and type of feeding. There is the possibility that the support will be held via "Skype" if the women prefer it.

<Activities for both groups (intervention and control)> Investigators will deliver written relevant information about the recommended alimentation of the women at postpartum as well as some ideas for physical activity. This technical information is derived from the literature and will be expressed in a simple and accessible way.

PHASE 3. FOLLOW-UP At a month postpartum, investigators will visit participants at home, both the control group and the intervention group, for information on breastfeeding practices. Also from the mother, a breast milk sample will be taken to determine the composition of fatty acids of it, a blood sample to determine C-Reactive Protein and also investigators will collect dietary information. Additionally, weight, length, and skinfold thickness of the baby will be taken. The project staff will be standardized for newborn anthropometric measurement, following the technique of Lohman.

Sample size and statistical power Investigators will study 200 obese pregnant women, 100 per study group. This sample size was calculated to detect a difference in the prevalence of exclusive breastfeeding (at one month postpartum) in 10 percent (12 to 22%), with a statistical power of 90%, a level of significance >0.05, a nonresponse rate of 50% and 15% of abandonment postpartum. To achieve the sample size, recruitment will be held for 5 months, hoping to incorporate to the study, at least, two women daily. This calculation was performed using information on the number of women who could meet the inclusion criteria of the study.

To achieve this sample size, investigators estimated to screen a total of 3,700 women in the primary care level health services in order to identify women who meet the inclusion criteria as described above.

According to similar studies, to calculate the number of women needed to get 200 women (100 in each group) investigators did as it follows:

All pregnant women attending health centers n= 3,700 It is expected that at least 34% of women have a body mass index (BMI)> 29 n= 1,258 It is expected that 40% meet inclusion criteria n= 503 Only 50% agree to participate n= 251 Approximately 80% give birth in the reference hospital n= 200

Data management Study participants will be assigned a unique identification number. A subject identification list will be created, including the subjects identification number, personal information and contact information of each subject participating in the study. Only the main investigator will have access to this list in order to make it possible to trace and identify an individual subject. This list will also help to carry out medical auditing. For all the analysis and data management, the identification number will be used in order to ensure confidentiality and privacy of the subjects.

Once data is collected by fieldworkers, the completed questionnaires will be brought to the headquarters of the study, where supervisors will check for potential mistakes or missing information. Investigators will use a case report form per participant, where a checklist of all information to be collected from them and the quality of it, will be recorded. The case report form will be filled out by the field supervisor every time is checking the file of each subject. The purpose of the case report form will be for monitoring the quality of the information collected, and to check that all the information is being collected on time.

Data entry will be performed continuously during the course of the study. Data will be entered in duplicate for quality control. In case there are missing data or errors in data collection, the fieldworkers will go back to participants and recover the information when possible. Regular backup of databases procedures will be conducted.

Statistical processing and analysis

Descriptive statistics (summary measures, according to variable type and measurement scale) including means, medians, standard errors and variances for each of the stages of data collection (baseline and follow-up), as applicable. To analyze baseline differences between the study groups, comparisons between groups will be made by the difference of proportions test for categorical variables and t tests for continuous variables. The statistics tests will include design information, adjusting the standard errors and applying a continuity correction.

For the analysis of sociodemographic information, a cluster analysis will be used to identify groups of interest considering some characteristics of women.

Analytical or inferential statistics (test to be applied by type of variable: if necessary, statistical hypotheses and test procedures).

To evaluate the effect of the intervention data will be analyzed as panel data comparisons of means and variances. ANOVA, ANCOVA MANOVA and for comparing the groups: analysis of variance with and without intervention between and within groups.

To evaluate the relationship between obesity and breastfeeding performance investigators will use regression models were conducted and sociodemographic and anthropometric of each of the participants and their children will be included.

On the other hand, regression models will be conducted to analyze the relationship between the composition of breast milk and the infant's growth at one month and at 12 months.

All the analysis will be done with intent to treatment.

Qualitative analysis For the analysis of the educational intervention, qualitative analysis will be carried out through satisfaction surveys and open-ended questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant Women <18 years old with a BMI >=28, and women <18 years old with a BMI >=27, utilizing their pre-pregnancy weight.
* Pregnant women within the second or early third trimester (week 20 through week 34 of gestation).

Exclusion Criteria:

* Pregnant women under 15 years old.
* Pregnant women diagnosed with HIV or AIDS, Hepatitis B and C, or the Human T lymphotropic virus. In the presence of these, women have the contraindication to feed their children with breast milk.
* Pregnant women with medical conditions that could interfere with breastfeeding, as severe infections transmitted through breast milk.
* Pregnant women with previous breast surgery (as breast reduction) because the lactiferous ducts end up damaged and may lead to poor or no milk production at all.
* Pregnant women that are taking medications that prevent carrying out breastfeeding.
* Pregnant women with a multiple pregnancy (in case of twins, the first born should be taken for the study).

Exit criteria:

* Newborns with less than 35 weeks of gestational age.
* Newborns dispatched to the neonatal intensive care unit (NICU) from the first day of life.
* Newborns who present major congenital malformations, severe enough to prevent the breastfeeding.

Elimination criteria:

* Newborns with hypertrophy (large for gestational age), because they may present hypoglycemia and therefore some should require to remain in fast even after starting oral feeding and especially on the first day of life.
* Newborns that enter to the Intermediate Care Unit for a neonatal or maternal adverse event even if the breastfeeding was already initiated.

Min Age: 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2016-07-14 (Actual); Primary Completion 2018-02-11 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Predominant breastfeeding prevalence | Within the first month of the child´s life
  Percentage of 1 month old (+- 1 week) infants who consume breastmilk as the principal source of nourishment; this includes expressed human milk from own mother. Predominantly breastfed means that it is possible that the infant had received the day prior to the interview, other source of feeding (water and water-based drinks, fruit juice) ritual fluids or ORS, drops or syrups (vitamins, minerals and medicines), and it excludes the consumption of infant formula.

SECONDARY OUTCOMES:
Exclusive breastfeeding prevalence | Within the first month of the child´s life
  Exclusively breastfed means that the infant received the day prior to the interview, no other food or drink, not even water, except breast milk (including milk expressed from own mother), but allows the infant to receive ORS, drops and syrups (vitamins, minerals and medicines).
Total duration of breastfeeding | During the 12 months of the child´s life
  The number of months the infants were breastfed; this variable will be evaluated up until the first 12 months of the infant's life.
WHO Child Growth Standards | At the first month and at the 12 months of infant´s life
  Comparison of the infants´s height for age, weight for height, weight for age and skinfolds, as compared to the 2008 WHO standards.

OTHER OUTCOMES:
Breastfeeding Self-Efficacy Scale-Short Form | Three times: Twice before delivery (once at baseline and again after the workshop), and a third occasion at the first month postpartum.
  Is the strength of the woman's belief in her's own ability to breastfeed her child.

CONTACTS AND LOCATIONS:
Overall Officials: Teresita González de Cosío, PhD., Study Chair — Universidad Iberoamericana, A.C.; Sonia L. Hernández Cordero, PhD., Principal Investigator — Universidad Iberoamericana, A.C.
Locations (1):
- Universidad Iberoamericana, A.C., Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No
The investigators do not plan to make IPD available

REFERENCES:
- [Background] Jevitt C, Hernandez I, Groer M. Lactation complicated by overweight and obesity: supporting the mother and newborn. J Midwifery Womens Health. 2007 Nov-Dec;52(6):606-13. doi: 10.1016/j.jmwh.2007.04.006. PMID 17983998
- [Background] Nommsen-Rivers LA, Chantry CJ, Peerson JM, Cohen RJ, Dewey KG. Delayed onset of lactogenesis among first-time mothers is related to maternal obesity and factors associated with ineffective breastfeeding. Am J Clin Nutr. 2010 Sep;92(3):574-84. doi: 10.3945/ajcn.2010.29192. Epub 2010 Jun 23. PMID 20573792
- [Background] Oddy WH, Li J, Landsborough L, Kendall GE, Henderson S, Downie J. The association of maternal overweight and obesity with breastfeeding duration. J Pediatr. 2006 Aug;149(2):185-91. doi: 10.1016/j.jpeds.2006.04.005. PMID 16887431
- [Background] Donath SM, Amir LH. Does maternal obesity adversely affect breastfeeding initiation and duration? J Paediatr Child Health. 2000 Oct;36(5):482-6. doi: 10.1046/j.1440-1754.2000.00562.x. PMID 11036806
- [Background] Li R, Jewell S, Grummer-Strawn L. Maternal obesity and breast-feeding practices. Am J Clin Nutr. 2003 Apr;77(4):931-6. doi: 10.1093/ajcn/77.4.931. PMID 12663294
- [Background] Wojcicki JM. Maternal prepregnancy body mass index and initiation and duration of breastfeeding: a review of the literature. J Womens Health (Larchmt). 2011 Mar;20(3):341-7. doi: 10.1089/jwh.2010.2248. PMID 21434834
- [Background] Hilson JA, Rasmussen KM, Kjolhede CL. Maternal obesity and breast-feeding success in a rural population of white women. Am J Clin Nutr. 1997 Dec;66(6):1371-8. doi: 10.1093/ajcn/66.6.1371. PMID 9394689
- [Background] León-Cava N, Lutter C, Ross Jay, Martin L. Quantifying the benefits of breastfeeding: a summary of the evidence. 2002; Available at: http://www1.paho.org/English/AD/FCH/BOB-Main.html.
- [Background] World Health Organization. Infant and young child feeding. Fact sheet 342. 2013; Available at http://www.who.int/mediacentre/factsheets/fs342/en/index.html. Revised on september of 2013.
- [Background] Eidelman AI. Breastfeeding and the use of human milk: an analysis of the American Academy of Pediatrics 2012 Breastfeeding Policy Statement. Breastfeed Med. 2012 Oct;7(5):323-4. doi: 10.1089/bfm.2012.0067. Epub 2012 Sep 4. No abstract available. PMID 22946888
- [Background] Gonzalez de Cosio T, Escobar-Zaragoza L, Gonzalez-Castell LD, Rivera-Dommarco JA. [Infant feeding practices and deterioration of breastfeeding in Mexico]. Salud Publica Mex. 2013;55 Suppl 2:S170-9. Spanish. PMID 24626693
- [Background] Barquera S, Campos-Nonato I, Hernandez-Barrera L, Pedroza A, Rivera-Dommarco JA. [Prevalence of obesity in Mexican adults 2000-2012]. Salud Publica Mex. 2013;55 Suppl 2:S151-60. Spanish. PMID 24626691
- [Background] Diet, nutrition, and the prevention of chronic diseases. Report of a WHO Study Group. World Health Organ Tech Rep Ser. 1990;797:1-204. No abstract available. PMID 2124402
- [Background] Obesity: preventing and managing the global epidemic. Report of a WHO consultation. World Health Organ Tech Rep Ser. 2000;894:i-xii, 1-253. PMID 11234459
- [Background] Astrup A, Dyerberg J, Selleck M, Stender S. Nutrition transition and its relationship to the development of obesity and related chronic diseases. Obes Rev. 2008 Mar;9 Suppl 1:48-52. doi: 10.1111/j.1467-789X.2007.00438.x. PMID 18307699
- [Background] Clark JM, Brancati FL. The challenge of obesity-related chronic diseases. J Gen Intern Med. 2000 Nov;15(11):828-9. doi: 10.1046/j.1525-1497.2000.00923.x. No abstract available. PMID 11119178
- [Background] Lawrence RA, Lawrence RM. Breastfeeding: A guide for the medical profession- 6th edition, Pensylvania. Elsevier MOSBY; 2005.
- [Background] Perez-Escamilla R, Curry L, Minhas D, Taylor L, Bradley E. Scaling up of breastfeeding promotion programs in low- and middle-income countries: the "breastfeeding gear" model. Adv Nutr. 2012 Nov 1;3(6):790-800. doi: 10.3945/an.112.002873. PMID 23153733
- [Background] Chapman DJ, Morel K, Anderson AK, Damio G, Perez-Escamilla R. Breastfeeding peer counseling: from efficacy through scale-up. J Hum Lact. 2010 Aug;26(3):314-26. doi: 10.1177/0890334410369481. PMID 20715336
- [Background] Chapman DJ, Morel K, Bermudez-Millan A, Young S, Damio G, Perez-Escamilla R. Breastfeeding education and support trial for overweight and obese women: a randomized trial. Pediatrics. 2013 Jan;131(1):e162-70. doi: 10.1542/peds.2012-0688. Epub 2012 Dec 3. PMID 23209111
- [Background] Rasmussen KM, Dieterich CM, Zelek ST, Altabet JD, Kjolhede CL. Interventions to increase the duration of breastfeeding in obese mothers: the Bassett Improving Breastfeeding Study. Breastfeed Med. 2011 Apr;6(2):69-75. doi: 10.1089/bfm.2010.0014. Epub 2010 Oct 19. PMID 20958105
- [Background] World Health Organization. Indicators for assessing infant and young child feeding practices. Part 3: country profiles. Geneva: WHO, 2008.
- [Background] Choque, R. Comunicación y educación para la promoción de la salud. FAS. Lima-Perú, 2005
- [Background] Organización Mundial para la Salud, Organización Panamericana de la Salud. Manual de comunicación social para programas de promoción de la salud de los adolescentes, 2001.
- [Background] US DEPARTMENT OF HEALTH & HUMAN SERVICES. Making health communication programs work. National Cancer Institute, 2001
- [Background] Organización Panamericana de la Salud. Herramientas de comunicación para el desarrollo de entornos saludables, 2006.
- [Background] Dyson L, McCormick F, Renfrew MJ. Interventions for promoting the initiation of breastfeeding. Cochrane Database Syst Rev. 2005 Apr 18;(2):CD001688. doi: 10.1002/14651858.CD001688.pub2. PMID 15846621
- [Background] Britton C, McCormick FM, Renfrew MJ, Wade A, King SE. Breastfeeding support, In: Cochrane Plus Library, 2008 Number 2. Oxford: Update Software Ltd. Available at: http://www.update-software.com. (The Cochrane Library, 2008 Issue 2. Chichester, UK: John Wiley & Sons, Ltd.).
- [Background] Bandura, A. Health promotion from the perspective of social cognitive theory. Psychol Health, 1998;13:623-649
- [Background] Clark MM, Abrams DB, Niaura RS, Eaton CA, Rossi JS. Self-efficacy in weight management. J Consult Clin Psychol. 1991 Oct;59(5):739-44. doi: 10.1037//0022-006x.59.5.739. PMID 1955608
- [Background] Eidman C. Enhancing Breastfeeding Self.Eficacy through Prenatal Education. Master of Arts in Nursing Theses, 2011;1-24.
- [Background] Baker JL, Gamborg M, Heitmann BL, Lissner L, Sorensen TI, Rasmussen KM. Breastfeeding reduces postpartum weight retention. Am J Clin Nutr. 2008 Dec;88(6):1543-51. doi: 10.3945/ajcn.2008.26379. PMID 19064514
- [Background] Dewey KG, Heinig MJ, Nommsen LA. Maternal weight-loss patterns during prolonged lactation. Am J Clin Nutr. 1993 Aug;58(2):162-6. doi: 10.1093/ajcn/58.2.162. PMID 8338042
- [Background] Gunderson EP, Jacobs DR Jr, Chiang V, Lewis CE, Feng J, Quesenberry CP Jr, Sidney S. Duration of lactation and incidence of the metabolic syndrome in women of reproductive age according to gestational diabetes mellitus status: a 20-Year prospective study in CARDIA (Coronary Artery Risk Development in Young Adults). Diabetes. 2010 Feb;59(2):495-504. doi: 10.2337/db09-1197. Epub 2009 Dec 3. PMID 19959762
- [Background] Ram KT, Bobby P, Hailpern SM, Lo JC, Schocken M, Skurnick J, Santoro N. Duration of lactation is associated with lower prevalence of the metabolic syndrome in midlife--SWAN, the study of women's health across the nation. Am J Obstet Gynecol. 2008 Mar;198(3):268.e1-6. doi: 10.1016/j.ajog.2007.11.044. Epub 2008 Jan 14. PMID 18191796
- [Background] Schwarz EB, Brown JS, Creasman JM, Stuebe A, McClure CK, Van Den Eeden SK, Thom D. Lactation and maternal risk of type 2 diabetes: a population-based study. Am J Med. 2010 Sep;123(9):863.e1-6. doi: 10.1016/j.amjmed.2010.03.016. PMID 20800156
- [Background] Stuebe AM, Rich-Edwards JW, Willett WC, Manson JE, Michels KB. Duration of lactation and incidence of type 2 diabetes. JAMA. 2005 Nov 23;294(20):2601-10. doi: 10.1001/jama.294.20.2601. PMID 16304074
- [Background] Kjos SL, Henry O, Lee RM, Buchanan TA, Mishell DR Jr. The effect of lactation on glucose and lipid metabolism in women with recent gestational diabetes. Obstet Gynecol. 1993 Sep;82(3):451-5. PMID 8355952
- [Background] Taylor JS, Kacmar JE, Nothnagle M, Lawrence RA. A systematic review of the literature associating breastfeeding with type 2 diabetes and gestational diabetes. J Am Coll Nutr. 2005 Oct;24(5):320-6. doi: 10.1080/07315724.2005.10719480. PMID 16192255
- [Background] Klein K, Bancher-Todesca D, Graf T, Garo F, Roth E, Kautzky-Willer A, Worda C. Concentration of free amino acids in human milk of women with gestational diabetes mellitus and healthy women. Breastfeed Med. 2013 Feb;8(1):111-5. doi: 10.1089/bfm.2011.0155. Epub 2012 Apr 27. PMID 22540840
- [Background] Ali MA, Strandvik B, Palme-Kilander C, Yngve A. Lower polyamine levels in breast milk of obese mothers compared to mothers with normal body weight. J Hum Nutr Diet. 2013 Jul;26 Suppl 1:164-70. doi: 10.1111/jhn.12097. Epub 2013 Apr 30. PMID 23627874
- [Background] Storck Lindholm E, Strandvik B, Altman D, Moller A, Palme Kilander C. Different fatty acid pattern in breast milk of obese compared to normal-weight mothers. Prostaglandins Leukot Essent Fatty Acids. 2013 Mar;88(3):211-7. doi: 10.1016/j.plefa.2012.11.007. Epub 2012 Dec 27. PMID 23273824
- [Background] Panagos P, Matthan N, Sen S. Effects of maternal obesity on breastmilk composition and infant growth. FASEB J April 2014 28:247
- [Background] Andreas NJ, Hyde MJ, Gale C, Parkinson JR, Jeffries S, Holmes E, Modi N. Effect of maternal body mass index on hormones in breast milk: a systematic review. PLoS One. 2014 Dec 23;9(12):e115043. doi: 10.1371/journal.pone.0115043. eCollection 2014. PMID 25536196
- [Background] Pedersen L, Lauritzen L, Brasholt M, Buhl T, Bisgaard H. Polyunsaturated fatty acid content of mother's milk is associated with childhood body composition. Pediatr Res. 2012 Dec;72(6):631-6. doi: 10.1038/pr.2012.127. Epub 2012 Sep 24. PMID 23007033
- [Background] Much D, Brunner S, Vollhardt C, Schmid D, Sedlmeier EM, Bruderl M, Heimberg E, Bartke N, Boehm G, Bader BL, Amann-Gassner U, Hauner H. Breast milk fatty acid profile in relation to infant growth and body composition: results from the INFAT study. Pediatr Res. 2013 Aug;74(2):230-7. doi: 10.1038/pr.2013.82. Epub 2013 May 28. PMID 23715519
- [Background] Dewey KG, Nommsen-Rivers LA, Heinig MJ, Cohen RJ. Risk factors for suboptimal infant breastfeeding behavior, delayed onset of lactation, and excess neonatal weight loss. Pediatrics. 2003 Sep;112(3 Pt 1):607-19. doi: 10.1542/peds.112.3.607. PMID 12949292
- [Background] Rasmussen KM, Kjolhede CL. Prepregnant overweight and obesity diminish the prolactin response to suckling in the first week postpartum. Pediatrics. 2004 May;113(5):e465-71. doi: 10.1542/peds.113.5.e465. PMID 15121990
- [Background] Esposito K, Pontillo A, Di Palo C, Giugliano G, Masella M, Marfella R, Giugliano D. Effect of weight loss and lifestyle changes on vascular inflammatory markers in obese women: a randomized trial. JAMA. 2003 Apr 9;289(14):1799-804. doi: 10.1001/jama.289.14.1799. PMID 12684358
- [Background] Hennigar S, Velasquez V and Kelleher S. Diet-induced obesity compromises lactation through zinc-mediated ER stress and autophagy, promoting premature involution. FASEB J April 2014; 28:910.4
- [Background] Nommsen-Rivers L, Glueck C, Huang B, Wang P, and Dolan L. Lactation sufficiency is predicted by fasting plasma glucose at 1 month postpartum (131.1) FASEB J April 2014;28:131.1
- [Background] Smith, L. J. Impact of birthing practices on breastfeeding, 2nd Ed. Sudbury, MA: Jones and Bartlett Publishers. (2010).
- [Background] Wagner EA, Chantry CJ, Dewey KG, Nommsen-Rivers LA. Breastfeeding concerns at 3 and 7 days postpartum and feeding status at 2 months. Pediatrics. 2013 Oct;132(4):e865-75. doi: 10.1542/peds.2013-0724. Epub 2013 Sep 23. PMID 24062375
- [Background] Matias SL, Nommsen-Rivers LA, Creed-Kanashiro H, Dewey KG. Risk factors for early lactation problems among Peruvian primiparous mothers. Matern Child Nutr. 2010 Apr;6(2):120-33. doi: 10.1111/j.1740-8709.2009.00195.x. PMID 20624209
- [Background] Geddes DT. Inside the lactating breast: the latest anatomy research. J Midwifery Womens Health. 2007 Nov-Dec;52(6):556-63. doi: 10.1016/j.jmwh.2007.05.004. PMID 17983992
- [Background] Lovelady CA. Is maternal obesity a cause of poor lactation performance. Nutr Rev. 2005 Oct;63(10):352-5. doi: 10.1111/j.1753-4887.2005.tb00113.x. PMID 16295148
- [Background] Evans A, Marinelli KA, Taylor JS; Academy of Breastfeeding Medicine. ABM clinical protocol #2: Guidelines for hospital discharge of the breastfeeding term newborn and mother: "The going home protocol," revised 2014. Breastfeed Med. 2014 Jan-Feb;9(1):3-8. doi: 10.1089/bfm.2014.9996. PMID 24456024
- [Background] Anstey EH and Jevitt C. Maternal Obesity and Breastfeeding A Review of the Evidence and Implications for Practice. Clinical Lactation, 2011;2-3:11-16
- [Background] Chambers JA, McInnes RJ, Hoddinott P, Alder EM. A systematic review of measures assessing mothers' knowledge, attitudes, confidence and satisfaction towards breastfeeding. Breastfeed Rev. 2007 Nov;15(3):17-25. PMID 18062138
- [Background] Fleiss JL, Levin B, Paik MC. Statistical Methods for Rates and Proportions. 3rd ed. New York: Wiley, 2003.
- [Background] Lohman T. Advances in body composition assessment. Human Kinetics. Champaign IL: Publishers; 1992.
- [Background] Ballard O, Morrow AL. Human milk composition: nutrients and bioactive factors. Pediatr Clin North Am. 2013 Feb;60(1):49-74. doi: 10.1016/j.pcl.2012.10.002. PMID 23178060
- [Background] Daly SE, Di Rosso A, Owens RA, Hartmann PE. Degree of breast emptying explains changes in the fat content, but not fatty acid composition, of human milk. Exp Physiol. 1993 Nov;78(6):741-55. doi: 10.1113/expphysiol.1993.sp003722. PMID 8311942
- [Background] Kent JC, Mitoulas LR, Cregan MD, Geddes DT, Larsson M, Doherty DA, Hartmann PE. Importance of vacuum for breastmilk expression. Breastfeed Med. 2008 Mar;3(1):11-9. doi: 10.1089/bfm.2007.0028. PMID 18333764
- [Background] Garcia-Lara NR, Escuder-Vieco D, Garcia-Algar O, De la Cruz J, Lora D, Pallas-Alonso C. Effect of freezing time on macronutrients and energy content of breastmilk. Breastfeed Med. 2012 Aug;7(4):295-301. doi: 10.1089/bfm.2011.0079. Epub 2011 Nov 2. PMID 22047109
- [Background] FOLCH J, LEES M, SLOANE STANLEY GH. A simple method for the isolation and purification of total lipides from animal tissues. J Biol Chem. 1957 May;226(1):497-509. No abstract available. PMID 13428781
- [Background] Lepage G, Roy CC. Direct transesterification of all classes of lipids in a one-step reaction. J Lipid Res. 1986 Jan;27(1):114-20. PMID 3958609
- [Background] Ledue TB, Weiner DL, Sipe JD, Poulin SE, Collins MF, Rifai N. Analytical evaluation of particle-enhanced immunonephelometric assays for C-reactive protein, serum amyloid A and mannose-binding protein in human serum. Ann Clin Biochem. 1998 Nov;35 ( Pt 6):745-53. doi: 10.1177/000456329803500607. PMID 9838988
- [Background] US Department of Health and Human Services. Food and Drug Administration. Review criteria for assessment of C-reactive protein (CRP), high sensitivity C-reactive protein (hsCRP) and cardiac C-reactive protein (cCRP) Assays. Document issued on: September 22, 2005. Available at: NK http://www.fda.gov/cdrh/oivd/guidance/1246.pdf
- [Background] Hartman AM, Brown CC, Palmgren J, Pietinen P, Verkasalo M, Myer D, Virtamo J. Variability in nutrient and food intakes among older middle-aged men. Implications for design of epidemiologic and validation studies using food recording. Am J Epidemiol. 1990 Nov;132(5):999-1012. doi: 10.1093/oxfordjournals.aje.a115743. PMID 2239915
- [Background] Manual de Instrumentos para la Evaluación Dietética. Guatemala: Instituto de Nutrición de Centro América y Panamá, 2006.
- [Background] National Institute of Public Health of Mexico. Food Composition Database. Unpublished document. 2013.
- [Background] Institute of Medicine. Energy. In: Dietary reference intakes for energy, carbohydrates, fiber, fat, protein and amino acids (macronutrients). Washington, DC: Institute of Medicine, The National Academies Press, 2005:107-264.
- [Background] Diet, nutrition and the prevention of chronic diseases. World Health Organ Tech Rep Ser. 2003;916:i-viii, 1-149, backcover. PMID 12768890